CLINICAL TRIAL: NCT06747494
Title: General Versus Spinal Anesthesia for Total Joint Arthroplasty: A Prospective Randomized Trial
Brief Title: General vs Spinal in Total Joint Arthroplasty (TJA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Victor Hugo Hernandez, Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20240978
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis
Keywords: Total joint arthroplasty; General anesthesia; Spinal anesthesia
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Anesthesia, General; Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia (Experimental): Participants in this group will receive general anesthesia for TJA for up to 2 hours.
  Interventions: Procedure: General Anesthesia
- Spinal Anesthesia (Experimental): Participants in this group will receive spinal anesthesia for TJA for up to 2 hours.
  Interventions: Procedure: Spinal Anesthesia

INTERVENTIONS:
Procedure: General Anesthesia — Participants will receive a one-time general anesthesia dose during the total joint arthroplasty procedure as per standard of care.
  Arms: General Anesthesia
Procedure: Spinal Anesthesia — Participants will receive a one-time spinal anesthesia dose during the total joint arthroplasty procedure as per standard of care.
  Arms: Spinal Anesthesia

SUMMARY:
The purpose of this research is to compare post-operative outcomes from patients undergoing TJA. The study team wants to learn about outcomes like length of hospital stay, post-operative pain scores, post-operative nausea, deep and superficial surgical site infection, periprosthetic fracture (a broken bone that occurs around an orthopaedic implant), implant dislocation, readmission rates, and revision rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary total hip or knee arthroplasty
* Subjects must be capable of providing informed consent
* English or Spanish speaking

Exclusion Criteria:

Patients with contraindications for spinal anesthesia such as:

* Prior lumbar surgery with hardware insertion
* Elevated intracranial pressure
* Infection at the site of the procedure
* Thrombocytopenia or coagulopathy
* Severe mitral and aortic stenosis and left ventricular outflow obstruction
* Severe spine pathology (spinal stenosis, spondylolisthesis, spondylosis) with radiculopathy and/or neurogenic claudication
* Preexisting neurological disease

Patients with contraindications for general anesthesia such as:

* Congestive heart failure
* Severe aortic stenosis
* Patient is unable/unwilling to consent
* Current pregnancy or women planning on becoming pregnant in the next year, and women who think they might be pregnant, or women who become pregnant during the study period will be removed from the study.
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2396 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Up to 72 hours.
  Will be measured in hours.
Change in Patient Pain Scores as measured by the Numeric Rating Pain Scale | Baseline (up to 1 hour after surgery), up to 24 hours.
  Score range from 0 to 10, higher score indicate higher pain scores.
Change in Patient Nausea Scores as measured by the Conditioning Scoring Criteria | Baseline (up to 1 hour after surgery), up to 24 hours.
  Score range from 0 to 9, higher score indicate higher nausea scores.
Prosthetic joint infection | Up to 90 days.
  Will be measured by the 2018 Musculoskeletal Infection Society criteria.
Superficial surgical site infection | Up to 90 days.
  Will be measured by the 2018 Musculoskeletal Infection Society criteria.
Number of periprosthetic fracture | Up to 90 days.
  Will be measured by the number of periprosthetic fracture.
Number of implant dislocation. | Up to 90 days.
  Will be measured by the number of implant dislocation.
Number of participants who are readmitted 90 days after surgery. | Up to 90 days.
  Will be measured by the number of participants who are readmitted 90 days after surgery.
Number of participants who receive revision surgery 90 days after surgery. | Up to 90 days.
  Will be measured by the number of participants who receive revision surgery 90 days after surgery.
Number of participant deaths. | Up to 90 days.
  Will be measured by the number of participants deaths.

SECONDARY OUTCOMES:
Length of surgery. | Up to 2 hours.
  Will be measured in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Victor H Hernandez, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No